CLINICAL TRIAL: NCT06112080
Title: Wearable Auscultation Device Validation in Children
Status: Terminated | Type: Observational
Why Stopped: The Principal Investigator is departing from the study site.
Sponsor: Strados Labs, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SL-LC01
Record Dates: First submitted 2023-10-23; First posted 2023-11-01 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2023-11

CONDITIONS: Asthma; Asthma in Children; Wheezing; Pediatric Asthma
MeSH Terms: conditions — Asthma; Respiratory Sounds

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Normal Breath Sound Cohort: 32 patients ages 4-10, 16 patients ages 11-17)
  * Admitted for a non-respiratory complaint
  * Normal breath sounds on screening examination
  Interventions: Device: RESP™ Biosensor
- Wheeze Cohort: (106 patients ages 4-10, 53 patients ages 11-17)
  * Admitted for pathologic process that may lead to wheezing (e.g., asthma)
  * Presence of wheeze on screening examination
  Interventions: Device: RESP™ Biosensor

INTERVENTIONS:
Device: RESP™ Biosensor — The RESP™ Biosensor will be placed on all participants for immediate capture and comparison of lung sounds.
  Other Names: Remote Electronic Stethoscope Platform

SUMMARY:
This observational clinical study is an evaluation of a diagnostic tool through comparison. Similar to a validation study, the output of the RESP device will be compared to physician auscultation, surrogated by having an attending pulmonologist listen to blinded recordings.

ELIGIBILITY:
Inclusion Criteria:

* Any child aged 4-17 years of age
* Admitted to Lurie Children's Hospital or the Emergency Department at Lurie
* Normal breath sounds cohort: (16 patients ages 4-10, 16 patients ages 11-17)

  * Admitted for a non-respiratory complaint
  * Normal breath sounds on screening examination
* Wheeze cohort: (53 patients ages 4-10, 53 patients ages 11-17)

  * Admitted for pathologic process that may lead to wheezing (e.g., asthma)
  * Presence of wheeze on screening examination

Exclusion Criteria:

* Children less than age 4, adults (age 18 and above)
* Patients in the ambulatory setting
* Unable to provide consent
* Intubated patients
* Unstable disease posing a threat to life
* Adhesive allergy

Ages: 4 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: pediatric subjects who present to Lurie Children's Hospital with or without wheezing.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2023-08-07 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Compare the output of the RESP Biosensor System to breath sound interpretation of an attending physician via collected recordings from stethoscope and completion of a comparison questionnaire | 12 months
  PI will compare Strados RESP portal output with concurrent recordings collected via Littmann 300 Stethoscope. A questionnaire will be used to record and determine similarities and differences between RESP output and Littmann output, ultimately validating the intended use. Spectrographic data and audio recordings obtained via auscultation will be collected respectively by the RESP device and a separate recording stethoscope (Littman CORE Digital Stethoscope) simultaneously. Demographic and clinical data will be collected and stored in REDcap.

SECONDARY OUTCOMES:
Tolerability and usability assessed utilizing The System Usibility Scale to evaluate attitudes towards the use and tolerance of the device by patients and caregivers | 12 months
  Assess the tolerability and usability of the Strados device by patients and caregivers utilizing the System Usability Scale will be used to evaluate subjects and caregivers attitudes towards the use and tolerance of the device. The System Usability Scale is a validated tool for evaluation of the usability and tolerability of a device or system by users. Then, subjects and caregivers will engage in a recorded interview using talk-aloud feedback. Recorded data will be transcribed and evaluated through quality analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided